CLINICAL TRIAL: NCT05055180
Title: Afterload Dependence of Right Ventricular Myocardial Remodeling and Intrinsic Right Ventricular Myocardial Function in Heart Failure With Preserved Ejection Fraction
Brief Title: Right Ventricular Function and Pulmonary Hypertension in HFpEF
Acronym: HFpEF-PHT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heart Center Leipzig - University Hospital (Other)
Collaborators: University Hospital Tuebingen (Other); University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: HFpEF-PHT 1.1
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biventricular myocardial tissue samples. Peripheral blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFpEF with pulmonary hypertension: Invasively diagnosed HFpEF and pulmonary hypertension according to current guidelines
  Interventions: Diagnostic Test: Invasive hemodynamics and myocardial biopsies
- HFpEF without pulmonary hypertension: Invasively diagnosed HFpEF without pulmonary hypertension according to current guidelines
  Interventions: Diagnostic Test: Invasive hemodynamics and myocardial biopsies
- Patients without HFpEF: Patients without invasive evidence of HFpEF
  Interventions: Diagnostic Test: Invasive hemodynamics and myocardial biopsies

INTERVENTIONS:
Diagnostic Test: Invasive hemodynamics and myocardial biopsies — Invasive hemodynamic characterization (biventricular pressure volume loop assessment) and biventricular myocardial biopsies

SUMMARY:
In patients with heart failure and preserved ejection fraction (HFpEF) right ventricular (RV) systolic and diastolic dysfunction are prognostically and functionally relevant factors but have mechanistically been neglected so far. In the present study alterations of intrinsic RV (systolic and diastolic) function, as assessed by invasive pressure volume loops, are examined in relation to tissue alterations on myocardial level and to the degree of RV afterload (pulmonary hypertension). Study aim is to gain insights into mechanisms contributing to the development of RV dysfunction and potentially identify new therapeutic targets.

ELIGIBILITY:
HFpEF

Inclusion Criteria:

* Clinical signs of heart failure
* Preserved Left ventricular (LV) Ejection Fraction (EF >= 50%)
* Structural Heart Diseases on echocardiogram/ N terminal-pro-brain natriuretic peptide > 125ng/l
* Elevated LV end-diastolic pressure at rest (>15mmHg) or during exertion (>=25mmHg)

No Heart Failure

Inclusion Criteria:

* No signs of heart failure
* Preserved Left ventricular (LV) Ejection Fraction (EF >= 50%)
* Normal LV end-diastolic pressure at rest (=<15mmHg) and during exertion (<25mmHg)

Exclusion Criteria:

* Significant coronary artery stenosis at time of catheterization
* Acute coronary syndrome or cerebral insult within 1 month of examination
* more than moderate valvular diseases
* pregnancy
* contraindication to cardiac magnetic resonance imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient general cardiology clinic
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Right ventricular systolic and diastolic function | Baseline
  Assessed with pressure volume loops analysis
Biventricular myocardial fibrosis | Baseline
  Assessed with histopathology
Phosphorylation of structural myocardial proteins | Baseline
  Assessed on myocardial biopsy specimen

SECONDARY OUTCOMES:
Functional capacity | Baseline
  6-Minute Walk Test / Spiroergometry
Myocardial fibrosis on cardiac magnetic resonance | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Center Leipzig at Leipzig University, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rommel KP, von Roeder M, Oberueck C, Latuscynski K, Besler C, Blazek S, Stiermaier T, Fengler K, Adams V, Sandri M, Linke A, Schuler G, Thiele H, Lurz P. Load-Independent Systolic and Diastolic Right Ventricular Function in Heart Failure With Preserved Ejection Fraction as Assessed by Resting and Handgrip Exercise Pressure-Volume Loops. Circ Heart Fail. 2018 Feb;11(2):e004121. doi: 10.1161/CIRCHEARTFAILURE.117.004121. PMID 29449367
- [Result] von Roeder M, Kowallick JT, Rommel KP, Blazek S, Besler C, Fengler K, Lotz J, Hasenfuss G, Lucke C, Gutberlet M, Thiele H, Schuster A, Lurz P. Right atrial-right ventricular coupling in heart failure with preserved ejection fraction. Clin Res Cardiol. 2020 Jan;109(1):54-66. doi: 10.1007/s00392-019-01484-0. Epub 2019 May 3. PMID 31053957